CLINICAL TRIAL: NCT05909202
Title: A Pilot Study of a Nature-Based Virtual Reality (VR) Intervention in Family Caregivers of Allogeneic Hematopoietic Stem Cell Transplant (HSCT) Recipients
Brief Title: A Nature-Based Virtual Reality (VR) Intervention in Family Caregivers of Allogeneic Hematopoietic Stem Cell Transplant (HSCT) Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10001636; 001636-CC
Record Dates: First submitted 2023-06-16; First posted 2023-06-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12-11

CONDITIONS: Neoplasm; Caregivers
Keywords: Hematopoietic Stem Cell Transplantation; Biobehavioral; Nature; Virtual Reality; Stress
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active VR Group (Experimental): Nature-based immersive VR program, completion of questionnaires, and saliva and blood sample submission.
  Interventions: Device: Active VR
- Sham VR Group (Sham Comparator): Nature-based non-immersive VR program, completion of questionnaires, and saliva and blood sample submission.
  Interventions: Device: Sham VR

INTERVENTIONS:
Device: Sham VR — Nature-based non-immersive VR program
  Arms: Sham VR Group
Device: Active VR — Nature-based immersive VR program
  Arms: Active VR Group

SUMMARY:
Background:

People who receive an allogeneic hematopoietic stem cell transplant (HSCT) require long-term care at home afterwards. Their caregivers often experience high levels of stress, which can lead to symptoms such as depression, anxiety, poor sleep, fatigue, and difficulties with concentration and memory.

Objective: To explore whether a nature-based immersive virtual reality (VR) program helps reduce stress in people who care for HSCT patients.

Eligibility:

People aged 18 and older who are primary caregivers of HSCT patients.

Design:

This is a two-phase study. Participants will be enrolled for 4 weeks. They will have 2 clinic visits.

Participants will have a physical exam at the beginning of the study. They will be asked to provide a saliva sample in Phase 1, and saliva and blood samples in Phase 2.

Participants will be given a VR headset. This is a device that looks like a pair of goggles worn over the eyes. They will be asked to wear the headset for 20 minutes per day. They will see 360 (Infinite) high-definition videos of nature and hear nature sounds.

Participants will record the time they spend using the VR headset in a daily diary. They will take surveys with questions about any stress and symptoms they feel once a week. This will take up to 5 minutes. Participants will have a short regular follow-up visit by phone one week after starting their participation.

At the end of the intervention study, participants will return for another physical exam. They will give saliva and/or blood samples again.

Researchers will also look at the medical records of the HSCT patients; the HSCT patients must consent to this.

DETAILED DESCRIPTION:
Study Description:

This is an interventional protocol to decrease stress and symptoms with a four-week nature-based VR intervention in family caregivers of allogeneic HSCT recipients. This study is a two-phase study: Phase I will be a single-arm pre-post design focused on assessing the feasibility and acceptability of the four-week nature-based immersive VR program. Phase II will be a prospective randomized controlled group design to examine the effectiveness of the four-week nature-based immersive VR program (Active VR) on stress and symptoms compared to a four-week nature-based non-immersive VR program (Sham VR) in the target population.

Objectives:

Phase I

Primary Objective: To evaluate the feasibility and acceptability of the nature-based immersive VR program in HSCT caregivers.

Secondary Objectives: To examine the level of perceived restorativeness, perceived stress, and symptoms (fatigue, sleep disturbance, depression, anxiety, cognitive impairment) in HSCT caregivers participating in the nature-based immersive VR program.

Exploratory Objectives: To examine relationships among variables including but not limited to perceived stress, symptoms, HSCT caregiver characteristics, HSCT recipient characteristics, and biomarkers.

Phase II

Primary Objective: To examine whether HSCT caregivers participating in Active VR demonstrate improved levels of perceived stress compared to those participating in Sham VR.

Secondary Objectives:

1. To examine whether HSCT caregivers participating in Active VR demonstrate improved levels of symptoms (fatigue, sleep disturbance, depression, anxiety, cognitive impairment) compared to those participating in Sham VR.
2. To examine the acceptability of Active and Sham VR programs in HSCT caregivers.

Exploratory Objectives: To examine relationships among variables including but not limited to perceived stress, symptoms, HSCT caregiver characteristics, HSCT recipient characteristics, and biomarkers.

Endpoints: Phase I

Primary Endpoints: Feasibility (recruitment, retention, and adherence rates) and acceptability (satisfaction, usability) measured at Time 4 (Day 28); acceptability (safety) from Time 0 (Baseline; Day 0) to Time 4

Secondary Endpoints: Perceived restorativeness measured at Time 4; changes in perceived stress from Time 0 to Time 4; changes in symptoms (fatigue, sleep disturbance, depression, anxiety, cognitive impairment) from Time 0 to Time 4

Phase II

Primary Endpoint: Changes in perceived stress from Time 0 to Time 4

Secondary Endpoints: Changes in symptoms (fatigue, sleep disturbance, depression, anxiety, cognitive impairment) from Time 0 to Time 4; acceptability (satisfaction, usability) measured at Time 4; acceptability (safety) from Time 0 to Time 4

ELIGIBILITY:
* INCLUSION CRITERIA:

Caregiver subjects

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Ability to understand and the willingness to sign a written informed consent document.
2. Age 18 years and older.
3. Serving as a primary caregiver* for an adult patient (18 years and older) planning to undergo their 1st allogeneic HSCT at the NIH Clinical Center during the four-week study period.
4. Ability to read, speak and understand English.
5. Access to necessary resources for participating in online survey (i.e., computer, laptop, tablet, smartphone, internet access).

   * If more than one caregiver is planned for the transplant recipient during the transplant phase, only one primary caregiver will be eligible to participate in the study. A primary caregiver is defined as someone who lives with or provides care regularly for the HSCT recipient during the 4-week study period. Caregivers will be categorized as to whether they are the sole caregiver versus one of the multiple caregivers.

HSCT recipient subjects

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Ability to understand and the willingness to sign a written informed consent document.
2. Age 18 years and older.
3. Planning to undergo their 1st allogeneic HSCT at the NIH Clinical Center during the four-week study period.
4. Ability to read, speak and understand English

EXCLUSION CRITERIA:

Caregiver subjects

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Serving as a paid caregiver for the patient.
2. Not agreeing to follow the study procedures.
3. Recent use of immersive VR programs for stress relief and/or entertainment (more than 2 days/week within the past 3 months). *
4. Participation in another stress-reduction type interventional study within the past 3 months.
5. Having a medical condition that is prone to frequent nausea or dizziness.
6. Current or past history of seizure, chronic migraines, epilepsy, claustrophobia, panic disorder, post-traumatic stress disorder, generalized anxiety disorder, major depressive disorder or other known severe neurological or mental health disorders.
7. Being sensitive to flashing light or motion.
8. Having a balance disorder such as vertigo and cybersickness.
9. Having another medical condition or injury that may prevent use of VR headset and/or VR software (e.g., visual or hearing problems, open sores, wounds, skin rash on face, or active infection).
10. Self-reported diagnosis of Opioid, Cocaine and/or Cannabis use disorder in the past year.

    * In Phase II, if a participant from Sham VR group personally uses immersive VR programs for stress relief and/or entertainment (more than 2 days/week) during the study period, the participant will be no longer eligible.

HSCT recipient subjects:

1. Not agreeing to follow the study procedures.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in perceived stress | 4 weeks
  The outcome will be used to assess the effects of the Active VR compared to the Sham VR.

SECONDARY OUTCOMES:
Changes in symptoms (fatigue, sleep disturbance, depression, anxiety, cognitive impairment), acceptability (satisfaction, usability), acceptability (safety) (Cross) (Cross) (Cross) | 4 weeks
  The outcome will be used to assess the effects of the Active VR compared to the Sham VR.

CONTACTS AND LOCATIONS:
Overall Officials: Lena J Lee, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee LJ, Son EH, Farmer N, Gerrard C, Tuason RT, Yang L, Kohn-Godbout J, Stephens C, Nahm ES, Smith L, Risch S, Wallen GR. Nature-based virtual reality intervention to manage stress in family caregivers of allogeneic hematopoietic stem cell transplant recipients: a two-phase pilot study protocol. Front Psychiatry. 2024 Mar 7;15:1295097. doi: 10.3389/fpsyt.2024.1295097. eCollection 2024. PMID 38516258
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001636-CC.html